CLINICAL TRIAL: NCT01155128
Title: Effects of an Exercise Program in Patients With Hypertensive Chronic Kidney Disease: a Randomized Clinical Trial
Brief Title: Effects of an Exercise Program in Patients With Hypertensive Chronic Kidney Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of Pelotas (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Principal Investigator, FRANKLIN CORREA BARCELLOS, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EPI-0001-FB
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Cardiovascular Disease; Chronic Kidney Disease; Chronic Renal Disease; Hypertension
Keywords: physical activity; exercise; sedentarism; chronic renal disease; failure renal chronic; proteinuria; progression; Renal Protective Effects of Exercise; quality of life changes with exercise in CKD; Endothelial progenitor cells in CKD; Chronic Kidney Disease and Ankle Brachial Index
MeSH Terms: conditions — Cardiovascular Diseases; Renal Insufficiency, Chronic; Hypertension; Motor Activity; Proteinuria; Disease Progression | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle interventions (Experimental): After recruitment of the participants and consented to participate those deemed eligible for inclusion completed baseline surveys will be randomly assigned to an intervention group and another control group that will receive the usual care
  Interventions: Behavioral: exercise aerobic
- lifestyle interventions (Placebo Comparator): After recruitment of the participants and consented to participate those deemed eligible for inclusion completed baseline surveys will be randomly assigned to an intervention group and another control group that will receive the usual care
  Interventions: Behavioral: exercise aerobic

INTERVENTIONS:
Behavioral: exercise aerobic — The intervention will consist of physical exercise sessions for approximately 60 minutes and two weekly sessions. The classes will consist of an initial part to exercises heating joint flexibility and lasting 10 minutes, a major part consists of aerobic exercise, lasting 20-30 minutes, and a piece of muscular endurance with exercises upper and lower limbs and abdomen, lasting 10-20 minutes. The intensity will be controlled through the Subjective Perception Scale Borg
  Other Names: aerobic exercise; exercício físico

SUMMARY:
Introduction: Chronic kidney disease (CKD) is now an important public health issue. While 0.1% of the population is on dialysis, approximately 4.5% of subjects have renal dysfunction (glomerular filtration rate <60 ml/min/1.73 m2). These patients have a high mortality of cardiovascular disease (CVD) with low quality of life and survival, despite high expenditure on their treatment. Hypertension (SAH) is both a cause and a complication of CKD. In addition, CKD and hypertension are risk factors for CVD. The nephropathy that are not on dialysis are less studied than those on dialysis. Strategies are needed to maintain renal function in these patients and mitigate the risk factors for CVD. A sedentary lifestyle can be an important determinant of morbidity of mortality. This study aims to determine the effect of exercise in patients with CKD not yet on dialysis.

Methodology: A randomized clinical trial in hypertensive patients with CRF. After recruitment of participants and completed baseline surveys, those eligible for inclusion and consented to participate in the study will be randomly assigned. We use the technique of randomization in blocks of fixed size of six persons.

Variables to be collected: demographic, socioeconomic, behavioral, anthropometric, blood pressure, laboratory tests (anemia, the lipid profile, blood glucose, inflammatory markers and number of peripheral endothelial progenitor cells) and quality of life. These patients will be re-interviewed in the middle period of the study (10 weeks) at the end of the intervention (20 weeks) and 10 weeks after the end of the intervention. The intervention group will participate in two weekly sessions of exercise.

Therefore, facing the epidemic of CKD, this study intends to fill the data gaps about the impact of physical activity in patients with CKD on dialysis.

DETAILED DESCRIPTION:
Eligibility:

Individuals hypertensives diagnosed with GFR between 15 and 59 ml/min./1.73m2

Will be excluded from the study following patients:

* Diabetes mellitus;
* Severe physical disability
* Acute myocardial infarction in the last six months;
* Uncontrolled hypertension (systolic pressure> 180 mmHg and / or diastolic pressure> 110 mmHg);
* Angina at rest (unstable) or triggered by exercise;
* Congestive heart failure (> class II New York Heart Association; table X);
* Cardiac arrhythmias (> Lown class II,> 30 premature beats per minute);
* Subjects with prior renal transplant or dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have hypertension diagnosed with Glomerular Filtration Rate from 15 to 59 ml/min./1.73m2 characterized, therefore, in stages 3 or 4 chronic kidney disease enrolled in Basic Health Units (BHU) in the urban area of Pelotas , RS.

Exclusion Criteria:

* Ia) Subjects diagnosed with diabetes mellitus; b) Patients with severe physical disability (lower limb amputation without prosthesis, orthopedic diseases that worsen with exercise); c) Individuals who have had acute myocardial infarction in the last six months; d) Subjects with hypertension at rest uncontrolled (systolic> 180 mmHg and / or diastolic pressure> 110 mmHg); e) Patients with angina at rest (unstable) or triggered by exercise; f) Individuals with congestive heart failure (> class II New York Heart Association; Table X); g) Patients with cardiac arrhythmias (> Lown class II,> 30 premature beats per minute); h) Individuals with peripheral vascular disease or moderate to severe; i) Subjects with prior renal transplant or dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-11 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Progression of renal disease | 30 th weeks
  randomized clinicals trials efficacy exercise in patients with chronic renal disease

SECONDARY OUTCOMES:
quality of life | 30th weeks
  assessing quality of life in patients with chronic kidney disease receiving conservative treatment: a randomized clinical trial
efficacy of physical exercise on blood pressure | 30 weeks
  same, patients pré-dialysis, randomized clinical trial
Effects of exercise on endothelial progenitor cells in pre-dialysis patients | 30 weeks
  same, endothelial progenitor cells in whole blood using flow cytometry (number)in pre-dialysis patients: randomized clinical trial
Ankle Brachial Pressure Index | 30 weeks
  same, association of Chronic Kidney Disease With the Spectrum of Ankle Brachial Index in patients pré-dialysis, randomized clinical trial
blood lipids | 30 weeks
  same, in patients pré-dialysis, randomized clinical tria

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Hallal, phd, Study Director — university federal de pelotas
Locations (1):
- University Federal of Pelotas, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Barcellos FC, Del Vecchio FB, Reges A, Mielke G, Santos IS, Umpierre D, Bohlke M, Hallal PC. Exercise in patients with hypertension and chronic kidney disease: a randomized controlled trial. J Hum Hypertens. 2018 Jun;32(6):397-407. doi: 10.1038/s41371-018-0055-0. Epub 2018 Apr 4. PMID 29615792
- See also: Center for Epidemiological Research — http://www.epidemio-ufpel.org.br